CLINICAL TRIAL: NCT06574087
Title: Determining the Frequency of Occurrence and Defining the Most Appropriate Screening Test for Anal Intraepithelial Neoplasia (AIN) in Patients With Human Papillomavirus (HPV) Related Gynecological Diseases.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PCK Marine Hospital in Gdynia (Other)
Collaborators: Medical University of Gdansk (Other); National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Michal Brzezinski, MD, PCK Marine Hospital in Gdynia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PCK01
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-08

CONDITIONS: HPV-Related Carcinoma; HPV Infection
Keywords: anal cancer; HPV; anal intraepithelial neoplasia
MeSH Terms: conditions — Papillomavirus Infections; Anus Neoplasms | interventions — Cytological Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HPV- related gynecological disease arm (Active Comparator)
  Interventions: Diagnostic Test: hrHPV test and cytology
- Placebo arm (Placebo Comparator)
  Interventions: Diagnostic Test: hrHPV test and cytology

INTERVENTIONS:
Diagnostic Test: hrHPV test and cytology — Perfomance of hrHPV test and cytology

SUMMARY:
The primary aim of the study is to determine the total risk of AIN in group of HPV-RGD survivors and additionally to establish an exact risk for each of HPV-related gynecological precancers/cancers. Moreover, the most appropriate screening test for HSIL(AIN) in this group of patients will be determined. It will be effectuated by performing two kinds of tests: hrHPV test for the 14 most common oncogenic HPV types and the liquid cytology from both the lower genital tract and anal canal with subsequent high resolution anoscopy (HRA) with potential biopsy/excision of suspected lesions and histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* HPV related gynecological disease confirmed in histo-pathological examination
* the posibility to obtain material from gynecological organ and from anal canal

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Anal intraepithelial neoplasm/ anal cancer | Just before surgery
  Number of Participants with anal intraepithelial neoplasm/ anal cancer among patients with HPV-related gynecological diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- PCK Marine Hospital in Gdynia, Gdynia, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided

REFERENCES:
- [Background] Brzezinski M, Stukan M. Anal Cancer and Anal Intraepithelial Neoplasia Risk among Patients Treated for HPV-Related Gynecological Diseases-A Systematic Review. J Clin Med. 2023 Jun 22;12(13):4216. doi: 10.3390/jcm12134216. PMID 37445251
- [Derived] Brzezinski M, Stukan M. Synchronous anal HPV Infection in Patients with HPV-Related Gynaecological Diseases: A Prospective Study. Infect Dis Ther. 2026 Jan;15(1):285-295. doi: 10.1007/s40121-025-01272-6. Epub 2025 Nov 26. PMID 41296233